CLINICAL TRIAL: NCT01213485
Title: Observational Cohort Study in Chronic Kidney Disease Patients on Dialysis Initiating Treatment With Mircera During the Correction and Maintenance Phase
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) in Patients With Chronic Kidney Disease on Dialysis (HORTENSIA)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22643
Record Dates: First submitted 2010-09-28; First posted 2010-10-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the course of treatment, the efficacy on anemia and the safety of Mircera (methoxy polyethylene glycol-epoetin beta) in patients with chronic kidney disease on dialysis. Eligible patients will be on either haemodialysis or peritoneal dialysis and treatment-naïve for or having had prior therapy with erythropoiesis stimulating agents (ESA). Data will be collected from each patient for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic kidney disease, on dialysis for > 3 months
* Treatment-naïve or previous treatment with ESA
* Initiation of treatment with Mircera for renal insufficiency associated anemia by decision of the treating physician

Exclusion Criteria:

* Participation in a clinical trial
* Anemia due to an associated malignant pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease on dialysis
Sampling Method: Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Haemoglobin levels | Month 6
Mircera therapy (dosage, schedule, mode of application) in the treatment of anemia in clinical practice | Month 6

SECONDARY OUTCOMES:
Change in haemoglobin/haematocrit | from baseline to Month 12
Biological parameters of anemia: transferrin saturation, serum ferritin, folates | 12 months
Efficacy of dialysis (Kt/V, urea levels) | 12 months
Safety: Incidence of adverse events | 12 months
Compliance (treatment modification or discontinuation) | 12 months
Quality of life: Short Form (SF-36) questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuilly-sur-Seine, France